CLINICAL TRIAL: NCT07068113
Title: Effects of Turkish Traditional Dances on Bone Mineral Density, Bone Turnover Markers, Balance, Aerobic Capacity and Quality of Life in Postmenopausal Osteopenic Women
Brief Title: Effects of Turkish Traditional Dances on Postmenopausal Osteopenic Women
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmet Faik Ulusoy, RESEARCH ASSISTANT, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AnkaraEtlik-FTR-AFU-01
Record Dates: First submitted 2025-07-04; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Osteopenic Women
Keywords: osteopenia; postmenopausal women; Turkish Dance; bone turnover markers; Bone Mineral Density
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXERCISE GROUP (Active Comparator): Patients are asked to do a home exercise program 3-5 days a week
  In addition to the exercises, they are asked to walk only 3 days a week, a total of at least 150 minutes per week
  Interventions: Other: EXERCISE GROUP
- DANCE GROUP (Active Comparator): A home exercise program will be done 3-5 days a week In addition to home exercises, patients will be asked to dance with a tempo determined by the study team before the study, lasting 30 minutes, accompanied by dance videos from various regions Before the dance, 10 minutes of WARM-UP EXERCISES will be asked, followed by 30 minutes of dance and 10 minutes of COOL-DOWN EXERCISES. Thus, it is aimed for you to dance at least 50 minutes at least 2 days a week. In addition, it is asked to walk at least 50 minutes at a pace once a week
  Interventions: Other: DANCE GROUP

INTERVENTIONS:
Other: DANCE GROUP — home exercise program + 50 min/week brisk walking + 100 min/week dance
  Arms: DANCE GROUP
Other: EXERCISE GROUP — home exercise program + 150 min/week brisk walking
  Arms: EXERCISE GROUP

SUMMARY:
The aim of this study is to evaluate the effects of regular Turkish regional dances, in addition to conventional exercises given with a home program, on the quality of life, balance, aerobic capacity, bone mineral density (femoral neck, total and lumbar L1-4 and L2-4 T scores) and bone turnover markers (Type 1 collagen C-telopeptide [CTX-1] and Serum Procollagen 1 N-terminal peptide [P1NP]) of postmenopausal osteopenic women aged 50-60 years. Our study also aims to evaluate the compliance of patients to the exercise programs given to postmenopausal osteopenic women.

-What is the effect of regular Turkish regional dances on balance, aerobic capacity, muscle strength, quality of life, Bone Mineral Densitometry and Bone Turnover Markers in postmenopausal osteopenic women?

DETAILED DESCRIPTION:
Patients who meet the criteria of our study will first be divided into 2 different groups by a closed envelope drawing method performed by a clinic secretary who is not involved in the study. Both groups will be asked to do a home exercise program 3-5 days a week. This home program will include the movements in the attached exercise sheets (Warm-up, Cool-down, Balance and Strengthening exercises, which were created from the sheets taken from https://theros.org.uk). It will be shown by the physiotherapist at the beginning of the study.

In addition to home exercises, participants in the first group will be asked to dance to dance videos from various regions, lasting 30 minutes, at a tempo determined by the study team before the study.

The dance videos will consist of rhythmic and tempo Turkish Regional Dances such as horon, Ankara Dance Tunes, and halay varieties. These videos have been uploaded to the ''Osteopeni folk dances'' YouTube channel and the links to these videos will be shared with the participants. (The videos will be closed to access during the study and only the video link owners will be able to access these videos. Links https://youtube.com/playlist?list=PLxRTiZv_4GGMtNYzIuGVsde6T_bzLt0V&si=W XRPO-GA1iWtGHuw, https://youtube.com/playlist?list=PLxRTiZv_4GGMVXcRx7uhntLdU4LtvmVC5&si =nvxk1VGbPia04xQF, https://youtube.com/playlist?list=PLxRTiZv_4GGMccS_iYDW3I_ ODCODEdTx&si=lD-7_fU1vWJ-ZQOn)

Before dancing, 10 minutes of warm-up, 30 minutes of dancing, and 10 minutes of cooling down exercises will be performed. It is planned that patients will dance at least 2 days a week for a minimum of 50 minutes. In addition, it is planned to reach a minimum of 150 minutes/week aerobic exercise target by having them walk briskly for at least 50 minutes once a week.

Participants in the 2nd group will not be prescribed dance, in addition to the home exercise program, they will be recommended to walk only 3 days a week, for a total of 150 minutes per week.

Participants in the 1st group will be given the FORM-1, and participants in the 2nd group will be given the FORM-2, and they will be asked to fill out these forms daily. The form-1 in will ask for the duration of the home exercises or Turkish folk dances that were performed that day. The form in FORM-2 will also ask for the duration of the home exercises that were performed that day. Both groups will also be given the FORM-3, and they will be asked to write down the complications that occurred during the daily exercise.

Only the study group (1st group) will be called monthly and issues such as whether the forms are filled out daily and compliance with the exercises will be discussed.

ELIGIBILITY:
Inclusion Criteria:

1. Being a postmenopausal woman between the ages of 50-60
2. Not having a known diagnosis of osteoporosis and not having taken any antiresorptive or anabolic agents before
3. Being diagnosed with osteopenia with DEXA taken in the last 6 months at Etlik City Hospital (femoral neck, femoral total L1-4 or L2-4 T score between -1 and -2.5)
4. Being literate
5. Having a 25-Hydroxy vitamin D level in the blood >20 µg/L
6. Having a phone that can be used for communication for oneself or one of the family members, as well as having a smart phone, tablet or computer that can be used to watch videos
7. Being willing to participate in the study

Exclusion Criteria:

1. Having a body mass index >30 kg/m2
2. Having an extremely sedentary lifestyle (International Physical Activity Scale-Inactive according to Short Form)
3. Presence of fragility fracture
4. Presence of malignancy
5. Presence of cardiovascular or respiratory system disease that will prevent exercise (unstable angina, uncontrolled atrial or ventricular arrhythmia, 3rd degree atrioventricular block, severe aortic stenosis, severe asthma-COPD)
6. Presence of current neurological disease that will prevent exercise (CVA, MS)
7. Presence of psychiatric disease that will prevent exercise or cause non-compliance in follow-ups
8. Presence of musculoskeletal system disease that will prevent exercise (Stage 3-4 osteoarthritis, severe spinal stenosis, severe radiculopathy, lumbar surgery within the last 1 year)
9. Presence of known inflammatory joint disease
10. Presence of advanced vision, hearing loss or vertigo etc. that will prevent the patient from doing exercises or regional dances. Having any disease that will disrupt harmony by causing balance problems
11. Using active estrogen or progesterone containing preparations
12. Presence of hyperthyroidism

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2026-02-19 (Estimated)

PRIMARY OUTCOMES:
Bone Turnover Markers(Type 1 collagen C-telopeptide) | three month
  Serum Type 1 collagen C-telopeptide (CTX-1) will be used for bone resorption.
Bone Turnover Markers(Serum Procollagen 1 N-terminal peptide) | three month
  Serum Procollagen 1 N-terminal peptide (P1NP) will be used for bone formation
Bone Mineral Density(Femoral Neck T scores) | six month
  In our study, femoral neck T scores bone mineral densities in g/cm2 will be noted with Dual-energy X-ray absorptiometry .Values obtained by bone mineral density (BMD) measurement are divided into diagnostic classification by the World Health Organization (WHO) as normal bone mass, low bone mass (osteopenia) and osteoporosis. Normal bone mass is above -1 standard deviation point relative to the mean bone mineral density of the young adult reference population (T score -1 and above). Osteopenia (low bone mass) is when the bone mineral density is below -1 standard deviation score and above -2.5 standard deviation points compared to the average bone mineral density of the young adult reference population (T score between -1 and -2.5). Osteoporosis is defined as bone mineral density below -2.5 standard deviation points compared to the average of the young adult reference population (T score below -2.5 points).
Bone Mineral Density(Femoral total T scores) | six month
  In our study, femoral total T scores and bone mineral densities in g/cm2 will be noted with Dual-energy X-ray absorptiometry.Values obtained by bone mineral density (BMD) measurement are divided into diagnostic classification by the World Health Organization (WHO) as normal bone mass, low bone mass (osteopenia) and osteoporosis. Normal bone mass is above -1 standard deviation point relative to the mean bone mineral density of the young adult reference population (T score -1 and above). Osteopenia (low bone mass) is when the bone mineral density is below -1 standard deviation score and above -2.5 standard deviation points compared to the average bone mineral density of the young adult reference population (T score between -1 and -2.5). Osteoporosis is defined as bone mineral density below -2.5 standard deviation points compared to the average of the young adult reference population (T score below -2.5 points).
bone mineral density(lumbar 1-4 Tscores) | six month
  In our study, lumbar 1-4 T scores bone mineral densities in g/cm2 will be noted with Dual-energy X-ray absorptiometry .Values obtained by bone mineral density (BMD) measurement are divided into diagnostic classification by the World Health Organization (WHO) as normal bone mass, low bone mass (osteopenia) and osteoporosis. Normal bone mass is above -1 standard deviation point relative to the mean bone mineral density of the young adult reference population (T score -1 and above). Osteopenia (low bone mass) is when the bone mineral density is below -1 standard deviation score and above -2.5 standard deviation points compared to the average bone mineral density of the young adult reference population (T score between -1 and -2.5). Osteoporosis is defined as bone mineral density below -2.5 standard deviation points compared to the average of the young adult reference population (T score below -2.5 points).
bone mineral density(lumbar 2-4 T scores) | six month
  In our study, lumbar 2-4 T scores bone mineral densities in g/cm2 will be noted with Dual-energy X-ray absorptiometry .Values obtained by bone mineral density (BMD) measurement are divided into diagnostic classification by the World Health Organization (WHO) as normal bone mass, low bone mass (osteopenia) and osteoporosis. Normal bone mass is above -1 standard deviation point relative to the mean bone mineral density of the young adult reference population (T score -1 and above). Osteopenia (low bone mass) is when the bone mineral density is below -1 standard deviation score and above -2.5 standard deviation points compared to the average bone mineral density of the young adult reference population (T score between -1 and -2.5). Osteoporosis is defined as bone mineral density below -2.5 standard deviation points compared to the average of the young adult reference population (T score below -2.5 points).

SECONDARY OUTCOMES:
BALANCE | three month
  Static and balance indicators will be checked with Tecnobody PK 252 isokinetic balance measurement system and additionally functional reach test will be noted.
muscle strength | three month
  Quadriceps muscle strength of the dominant side will be checked with the Lafayette device.
aerobic capacity | three month
  Aerobic capacity will be measured with a 6-minute walk test
quality of life measurement | three month
  Quality of life will be measured with the Quality Of Life Questionnaire of the European Foundation for Osteoporosis-41 (QUALEFFO-41) Scale.
  QUALEFFO-41 consists of 5 subscales examining the five dimensions of health, such as pain (5 items), physical function (17 items), social function (7 items), general health assessment (3 items) and mental function (9 items). Validity and reliability for Turkish was done by Koçyiğit and his colleagues.
  The answers to the questions in the QUALEFFO-41 scale are scored from 1 (healthy) to 5 (unhealthy) in the order of options. The section score and total score are calculated by transferring the scores to a measurement out of 100. For each subgroup and total result in the scale, a score of 0 indicates the best health status, while a score of 100 indicates the worst health status

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik Ciy Hospital, Ankara, yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No